CLINICAL TRIAL: NCT01244711
Title: An Open-label Pilot Study to Examine the Value of Substituting Quetiapine for Benzodiazepines in Treatment-refractory Patients With Unipolar Depression or Generalized Anxiety Disorder and Chronic Benzodiazepine Use
Brief Title: Open-Label Pilot Study to Examine the Value of Substituting Quetiapine for Benzodiazepines
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Terminated: recruiting or enrolling participants has halted prematurely
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRUSQUET0483
Record Dates: First submitted 2010-11-18; First posted 2010-11-19 (Estimated); Results first posted 2015-03-06 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-03

CONDITIONS: Major Depression; Generalized Anxiety Disorder
Keywords: Major Depression; Generalized Anxiety Disorder; Benzodiazepine; Quetiapine
MeSH Terms: conditions — Depressive Disorder, Major; Generalized Anxiety Disorder | interventions — Quetiapine Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Quetiapine (Experimental): Dosing will begin with Seroquel-XR 50 mg. at bedtime and will escalate weekly to Seroquel-XR 100mg., Seroquel-XR 200mg. and Seroquel-XR 300 mg depending on clinical response and side effects.
  Interventions: Drug: quetiapine

INTERVENTIONS:
Drug: quetiapine — Dosing will begin with Seroquel-XR 50 mg. at bedtime and will escalate weekly to Seroquel-XR 100mg., Seroquel-XR 200mg. and Seroquel-XR 300 mg depending on clinical response and side effects.
  Other Names: Seroquel-XR

SUMMARY:
The hypothesis of this study is that symptoms of anxiety, depression and insomnia; and indices of psychosocial function will all improve, while BZ use will decrease significantly during a twelve-week trial period of substituting quetiapine for benzodiazepines.

DETAILED DESCRIPTION:
1.1 Background Numerous patients having depression or anxiety appear to use benzodiazepines chronically and respond incompletely to conventional antidepressants. These patients are more likely to request or incur frequent changes of medication because of non-response, incomplete response or intolerance. The hypothesis of this study is that symptoms of anxiety, depression and insomnia; and indices of psychosocial function will all improve, while BZ use will decrease significantly during a twelve-week trial period of substituting quetiapine for benzodiazepines.

1.2 Rationale for this study The scientific rationale for this derives from a combination of clinical observation and a review of the literature. Anecdotal clinical experience with numerous patients having depression or anxiety suggested to me that patients with chronic benzodiazepine use were less likely to respond or remit with conventional antidepressants and more likely to request or incur frequent changes of medication because of non-response, incomplete response or intolerance. Although most of these patients were not drug abusers and the doses they took were within ranges recommended in the package inserts for these drugs (e.g., 5-20mg/ day of diazepam or equivalent), they were "dependent" in the sense that they took the BZ daily or almost daily, would not give it up in spite of "good responses" (although often with residual symptoms of anxiety or insomnia) to antidepressants or mood stabilizers, and were determined to get their prescription refills on time and often upset if they could not. I hypothesized that chronic benzodiazepine use created circadian or ultradian cycles of sedation, which might be experienced as fatigue or amotivation, and withdrawal, which might be experienced as anxiety or insomnia. Patients often tinkered with the doses and timing of the doses in an attempt to smooth out these cycles. The current study will determine whether symptoms of anxiety, depression and insomnia; and indices of psychosocial function improve, while BZ use decreases during a twelve-week trial period of substituting quetiapine for benzodiazepines. This would be a proof of concept study in a unique subpopulation with MDD or GAD.

2. STUDY OBJECTIVES 2.1 Primary objective For MDD:The primary efficacy measures will be change from baseline to endpoint in the MADRAS and the change in mean daily benzodiazepine dose in diazepam equivalents during the past week.

For GAD: The primary efficacy measures will be change from baseline to endpoint in the HAM-A and the change in mean daily benzodiazepine dose in diazepam equivalents during the past week.

2.2 Secondary objectives Secondary efficacy measures will include response and remission rates and self-rated scales of symptoms and psychosocial function (the IDS-SR for depressive symptoms, the SAS-SR for social/vocational function and the Q-LES-Q for quality of life).

3. STUDY PLAN AND PROCEDURES 3.1 Overall study design and study plan Subjects will be followed to assure a stable regimen of antidepressant medications and BZ for at least 8 weeks. Patients will then be treated with flexible doses of quetiapine-ER up to 300mg/day for 8 weeks. Dosing will begin with Seroquel 50 mg. at bedtime and will escalate weekly to Seroquel 100mg., Seroquel-XR 200mg. and Seroquel-XR 300 mg depending on clinical response and side effects. BZ doses will be gradually tapered at the equivalent of 5mg/day/week of diazepam equivalents where possible. This is not a forced titration schedule.

3.2 Rationale for study design, doses and control groups The design is an open-label, proof of concept study. The dosing is based on my prior clinical experience with this patient population. There are no control groups.

3.4 Treatments 3.4.1 Identity of investigational product and comparators Seroquel-XR 50 mg., Seroquel-XR100mg., Seroquel-XR 200mg. and Seroquel-XR 300 mg.

3.4.2 Doses and treatment regimens Dosing will begin with Seroquel-XR 50 mg. at bedtime and will escalate weekly to Seroquel-XR 100mg., Seroquel-XR 200mg. and Seroquel-XR 300 mg depending on clinical response and side effects.

3.5 Pre-study, concomitant and post-study treatment(s)

Prohibited medication during the study:

* Potent cytochrome P450 inhibitors (including but not limited to ketoconazole, itraconazole, fluconazole, erythromycin, clarithromycin, troleandomycin, indinavir, nelfinavir, ritonavir, fluvoxamine and saquinavir)
* potent cytochrome P450 inducers (including but not limited to phenytoin, carbamazepine, barbiturates, rifampin, St. John's Wort, and glucocorticoids)
* Any psychotropic besides quetiapine, antidepressant or benzodiazepine.

Other medication, which is considered necessary for the subject's safety and well-being, may be given at the discretion of the investigator(s). The administration of all medication (including investigational products) must be recorded in the appropriately.

4. OUTCOME AND VARIABLES 4.1 Primary Variable For MDD: The primary efficacy measures will be change from baseline to endpoint in the MADRAS and the change in mean daily benzodiazepine dose in diazepam equivalents during the past week.

For GAD: The primary efficacy measures will be change from baseline to endpoint in the HAM-A and the change in mean daily benzodiazepine dose in diazepam equivalents during the past week.

4.2 Secondary Variables Secondary efficacy measures will include response and remission rates and self-rated scales of symptoms and psychosocial function (the IDS-SR for depressive symptoms, the SAS-SR for social/vocational function and the Q-LES-Q for quality of life).

4.3 Efficacy Variable(s) For MDD: The primary efficacy measures will be change from baseline to endpoint in the MADRAS and the change in mean daily benzodiazepine dose in diazepam equivalents during the past week.

For GAD: The primary efficacy measures will be change from baseline to endpoint in the HAM-A and the change in mean daily benzodiazepine dose in diazepam equivalents during the past week.

An overdose is not regarded as an AE. All symptoms associated with the overdose should however be reported as AEs. For further information regarding overdose, see section 11.2.

Pregnancy in itself is not regarded as an AE unless there is a suspicion that an investigational product may have interfered with the effectiveness of a contraceptive medication. For further details regarding pregnancy, see section 11.3.

4.4.1.3 Reporting of serious adverse events Investigators and other site personnel must inform the FDA, via a Medwatch form, of any unexpected and possibly Study Drug-related serious adverse events (SAEs) according to the FDA reporting requirement timelines. The Investigator must also inform appropriate AstraZeneca representatives of any SAE that occurs in the course of the study within one day (ie, immediately but no later than the end of the next business day) of when he or she becomes aware of it. The investigator must also report follow-up information on SAEs within one day. A copy of the MedWatch report must be faxed to AstraZeneca at the time the event is reported to the FDA. Reporting to the FDA is recommended regardless of whether an IND is required for the study.

Additionally, the Investigator shall provide AstraZeneca with a report of all other SAEs that did not qualify for expedited reporting to the FDA (e.g., considered to be expected and/or not related) on at least a quarterly basis in order for AstraZeneca to meet its regulatory reporting obligations.

If the Study is blinded, the Institution shall provide AstraZeneca with the code break information with the initial SAE report or a copy of the randomization schedule at the start of the Study, so that AstraZeneca may un-blind SAE reports to the extent necessary to meet global regulatory reporting requirements.

A complete written SAE report must be sent with a cover page indicating the following:

Drug Name (Seroquel); this is an Investigator Sponsored Study (ISS) Research (Protocol) and AstraZeneca Tracking Number [IRUSQUET0483] Principal Investigator's IND number assigned by the FDA (if applicable) Principal Investigator's full name and address Unblinding information (if applicable) Send by way of fax to Seroquel ISS Safety Representative (302) 885-3043

If a non-serious AE becomes serious, this and other relevant follow-up information must also be provided to AstraZeneca and the FDA within 1 day as described above. All SAEs have to be reported to AstraZeneca, whether or not considered causally related to the investigational product. All SAEs will be documented. The investigator is responsible for informing the IRB and/or the Regulatory Authority of the SAE as per local requirements.

4.4.2 Other safety measurements and variables Safety assessments will include vital signs at each visit and hematology, chemistries, pregnancy testing and urine drug screening prior to and at the end of treatment.

4.5 Volume of blood sampling and handling of biological samples The total volume of blood that will be drawn from each subject in this study is as follows: 30 cc 5. DATA MANAGEMENT We will develop standardized paper forms for collecting all data needed on study subjects including eligibility, demographic and other baseline data, sequential clinical assessments, dosing information, side effects, and outcome measures. all data required to explore the study hypotheses will be collected and entered into a database in the appropriate format for data analysis.

6. STATISTICAL METHODS AND DETERMINATION OF SAMPLE SIZE 6.1 Description of analysis populations All analyses will be conducted on the intention-to-treat population. 6.2 Method of statistical analysis The Wilcoxon signed-rank test will be applied to the mean scores available at weeks 0 vs. endpoint for the primary outcome measures: MADRS, HAM-A & daily BZ dose, and for the secondary outcome measures IDS-SR, SAS-SR and Q-LES-Q respectively to test the questions of whether there is a difference from pre- to post-quetiapine treatment. Separate tests will be conducted for the two diagnostic groups (MDD and GAD), but there is no intent to compare the two.

The proportions of a priori-defined responders and remitters during the study will be reported in descriptive statistics.

6.3 Determination of sample size NA The N of 20 per group is dictated by budget and feasibility considerations. This is a pilot study with no control or comparison groups. Under a 2-tailed α value of .05, we will have the power to detect a large effect size.

ELIGIBILITY:
Inclusion Criteria:

For inclusion in the study subjects must fulfil all of the following criteria:

1. Provision of written informed consent
2. A diagnosis of a current major depressive episode (n =20) or generalized anxiety disorder (n = 20) of at least 4 weeks duration, as defined by Diagnostic and Statistical Manual of Mental Disorders- Fourth Edition (DSM-IV) and assessed on the SCID. Subjects may be included if they meet criteria for double depression, i.e., current major depression with antecedent dysthymic disorder, major depression in partial remission or bipolar depression. MDD subjects must have a 24 item Hamilton Depression Rating Scale Score (HAM-D) at intake >/= 20. GAD subjects must have a Hamilton Anxiety Rating Scale Score (HAM-A) at intake >/= 20. Patients who meet criteria for current GAD only during a current episode of MDD will be considered to have MDD, according to DSM-IV convention.
3. Females and/or males aged 18-65 years
4. Female patients of childbearing potential must be using a reliable method of contraception and have a negative urine human chorionic gonadotropin (HCG) test at enrolment
5. Able to understand and comply with the requirements of the study
6. All subjects must report BZ use more days than not persistent for more than 6 months and a stable regimen of mood stabilizers and/or antidepressant medication for at least 8 weeks.

   -

Exclusion Criteria:

* Any of the following is regarded as a criterion for exclusion from the study:

  1. Pregnancy or lactation
  2. Any DSM-IV Axis I disorder not defined in the inclusion criteria
  3. Axis II diagnosis of antisocial, schizotypal or severe borderline personality disorder(defined as patients who are high risk for being unable to complete the study due to hospitalization, suicide attempts, significant self-mutilation, or other self-injurious or destructive behavior).
  4. Patients who, in the opinion of the investigator, pose an imminent risk of suicide or a danger to self or others
  5. Known intolerance or lack of response to quetiapine fumarate as judged by the investigator
  6. Use of any of the following cytochrome P450 3A4 inhibitors in the 14 days preceding enrolment including but not limited to: ketoconazole, itraconazole, fluconazole, erythromycin, clarithromycin, troleandomycin, indinavir, nelfinavir, ritonavir, fluvoxamine and saquinavir
  7. Use of any of the following cytochrome P450 inducers in the 14 days preceding enrollment including but not limited to: phenytoin, carbamazepine, barbiturates, rifampin, St. John's Wort, and glucocorticoids
  8. Administration of a depot antipsychotic injection within one dosing interval (for the depot) before randomisation
  9. Substance or alcohol dependence at enrolment (except dependence in full remission, and except for caffeine or nicotine dependence), as defined by DSM-IV criteria
  10. Opiates, amphetamine, barbiturate, cocaine, cannabis, or hallucinogen abuse by DSM-IV criteria within 4 weeks prior to enrolment
  11. Medical conditions that would affect absorption, distribution, metabolism, or excretion of study treatment
  12. Unstable or inadequately treated medical illness (e.g. diabetes, angina pectoris, hypertension) as judged by the investigator
  13. Involvement in the planning and conduct of the study
  14. Previous enrolment or randomisation of treatment in the present study.
  15. Participation in another drug trial within 4 weeks prior enrolment into this study or longer in accordance with local requirements

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2008-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: james h kocsis, md, Principal Investigator — weill cornell mc
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Quetiapine
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Quetiapine
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 48 [48 to 48]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Montgomery Asberg Depression Rating Scale (MADRS)
Description: For MDD: The primary efficacy measures will be change from baseline to endpoint in the MADRS and the change in mean daily benzodiazepine dose in diazepam equivalents during the past week. Range is 0 (least severe) to 50 (most severe).
Time Frame: 12 weeks
Population: Change in total score on the MADRS from baseline to final visit
Measure: Number; unit: units on a scale
Arm/Group | Quetiapine
Number analyzed (Participants) | 1
units on a scale | -12

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Quetiapine
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No